CLINICAL TRIAL: NCT00014222
Title: A Phase III Adjuvant Trial Of Sequenced EC + Filgrastim + Epoetin Alfa Followed By Paclitaxel Versus Sequenced AC Followed By Paclitaxel Versus CEF As Therapy For Premenopausal Women And Early Postmenopausal Women Who Have Had Potentially Curative Surgery For Node Positive Or High Risk Node Negative Breast Cancer
Brief Title: Combination Chemotherapy With or Without Colony-stimulating Factors in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA21; CAN-NCIC-MA21 (Registry Identifier: PDQ Identifier); AMGEN-CAN-NCIC-MA21 (Other: Drug Industry); NCCTG-CAN-NCIC-MA21 (Other: Participating group identifier); BMS-CAN-NCIC-MA21 (Other: Drug Industry); JANSSEN-ORTHO-CAN-NCIC-MA21 (Other: Drug Industry); PFIZER-CAN-NCIC-MA21 (Other: Drug Industry); SWOG-CAN-NCIC-MA21 (Other: Participating group identifier); CDR0000068520 (Other: PDQ); CALGB-CAN-NCIC-MA21 (Other: Participating group)
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epoetin Alfa; Filgrastim; Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: CEF (Active Comparator): 6 cycles - q 28 days (6 months) - Cyclophosphamide 75 mg/m2 - po - Days 1-14 - Epirubicin 60 mg/m2 - IV - Days 1 and 8 - 5 Fluorouracil: 500mg/m2 - IV - Days 1 and 8 + Continuous Antibiotic Prophylaxis with Cotrimoxazole 960 mg (i.e.2x480 mg tablets) po-bid or Ciprofloxacin 500 mg - po-bid
  Interventions: Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil
- Arm 2: EC/T (Active Comparator): 6 cycles - q 14 days (3 months) - Epirubicin 120 mg/m2 - IV - Day 1 - Cyclophosphamide 830 mg/m2 - IV - Day 1 - Filgrastim 5μg/kg/d - SC - Days 2 - 13 + Epoetin Alfa 40,000 IU - SC - once weekly (to begin within 1 week after start of protocol therapy as needed) 21 days from last administration of EC (EC/T) 4 cycles - q 21 days (3 months) - Adriamycin 60 mg/m2 - IV - Day 1 - Cyclophosphamide 600 mg/m2 - IV - Day 1 - 21 days from last administration of AC 4 cycles - q 21 days (3 months) - Paclitaxel 175 mg/m2 IV 3 hour infusion
  Interventions: Biological: epoetin alfa; Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel
- Arm 3: AC/T (Active Comparator): 4 cycles - q 21 days (3 months) - Adriamycin 60 mg/m2 - IV - Day 1 - Cyclophosphamide 600 mg/m2 - IV - Day 1 21 days from last administration of AC 4 cycles - q 21 days (3 months) - Paclitaxel 175 mg/m2 IV 3 hour infusion
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Biological: epoetin alfa — 40,000 IU
  Arms: Arm 2: EC/T
Biological: filgrastim — 5 mg/kg/d - days 2-13
  Arms: Arm 2: EC/T
Drug: cyclophosphamide — 75, 600 and 830 mg/m2
Drug: doxorubicin hydrochloride — 60 mg/m2
  Arms: Arm 2: EC/T; Arm 3: AC/T
Drug: epirubicin hydrochloride — 60 mg/m2
  Arms: Arm 1: CEF
Drug: fluorouracil — 500mg/m2
  Arms: Arm 1: CEF
Drug: paclitaxel — 175 mg/m2
  Arms: Arm 2: EC/T; Arm 3: AC/T

SUMMARY:
RATIONALE:

1. . To compare the effects on breast cancer of three different combinations of drugs which are commonly used to treat this disease.
2. . It is not yet known which treatment regimen is most effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy given with or without epoetin alfa in treating women who have undergone surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival of premenopausal or early postmenopausal women with previously resected node positive or high-risk node negative stage I-IIIB breast cancer treated with cyclophosphamide, epirubicin, and fluorouracil vs cyclophosphamide, epirubicin, filgrastim (G-CSF), and epoetin alfa followed by paclitaxel vs cyclophosphamide and doxorubicin followed by paclitaxel.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the rate of toxic effects of these regimens in this patient population.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of positive nodes (0 vs 1-3 vs 4-10 vs more than 10), type of prior surgery (total vs partial mastectomy), and estrogen receptor status (positive vs negative). Patients are randomized to one of three treatment arms.

* Arm I: Patients receive epirubicin IV and fluorouracil IV on days 1 and 8 and oral cyclophosphamide on days 1-14. Treatment repeats every 28 days for 6 courses.
* Arm II: Patients receive epirubicin IV and cyclophosphamide IV on day 1 and filgrastim (G-CSF) subcutaneously (SC) on days 2-13. Patients with a hemoglobin < 13.0 g/dL also receive epoetin alfa SC once weekly beginning within 1 week after the start of therapy and continuing as needed. Treatment repeats every 14 days for 6 courses. Beginning 21 days after completion of epirubicin and cyclophosphamide, patients receive paclitaxel IV over 3 hours on day 1 and G-CSF and epoetin alfa as above. Treatment repeats every 21 days for 4 courses.
* Arm III: Patients receive doxorubicin IV over 15 minutes and cyclophosphamide IV over 15 minutes on day 1. Treatment repeats every 21 days for 4 courses. Beginning 21 days after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel as in arm II. Treatment in all arms continues in the absence of disease progression or unacceptable toxicity.

All receptor positive patients receive oral tamoxifen or anastrozole (if tamoxifen is contraindicated) for 5 years after completion of chemotherapy.

Quality of life is assessed at baseline, day 1 of cycles 2, 3 4 and 6 (arm I), days 1 of cycles 3 and and day 1 of cycles 1 and 4 of paclitaxel (arm II), day 1 of cycles 2 and 3, day 1 of cycles 1 and 4 of paclitaxel, (arm III), 9 months, 12 months, and then annually thereafter until 5 years

Patients are followed at 9 months, 12 months, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,100 patients (700 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast that is potentially curable

  * T0-4 (dermal involvement on pathology assessment only), N0-2, M0
  * No clinical T4 disease
* Previously treated with one of the following:

  * Total mastectomy and level II axillary node dissection
  * Partial mastectomy and level II axillary node dissection with planned breast radiotherapy after completion of adjuvant chemotherapy regimen*
  * Patients with a positive sentinel node biopsy must undergo level II axillary node dissection or sufficient nodal sampling
  * If microscopic residual in situ or invasive disease is present at total or partial mastectomy margins, planned radiotherapy must also include a boost to the tumor bed
* No residual tumor in the axilla after dissection
* Axillary node positive

  * Negative nodes allowed if the tumor is ≥ 1 cm and 1 or more of the following criteria defining high-risk node-negative disease are met:

    * Histological grade III or,
    * Estrogen receptor negative or,
    * Lymphatic/vascular invasion
* Hormone receptor status:

  * Estrogen receptor status known

PATIENT CHARACTERISTICS:

Age:

* 60 and under

Sex:

* Female

Menopausal status:

* Pre- or postmenopausal

Performance status:

* ECOG 0-2

Life expectancy:

* At least 5 years

Hematopoietic:

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)

Renal:

* Creatinine ≤ 1.5 times ULN

Cardiovascular:

* LVEF ≥ limit of normal by MUGA or echocardiogram
* No arrhythmia requiring ongoing treatment
* No congestive heart failure
* No documented coronary artery disease

Other:

* No other malignancy except:

  * Adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
  * Ductal or lobular carcinoma in situ that has been curatively treated by surgery alone
  * Other prior malignancies (except breast cancer) curatively treated more than 5 years prior to study entry
* No serious underlying medical illness or psychiatric or addictive disorder that would preclude study compliance
* No known hypersensitivity to E. coli-derived products, mammalian-cell derived products, or any study agents
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for breast cancer
* No concurrent pegfilgrastim or darbepoetin alfa (Arm II)

  * Allowed on arms 1 and 3 if medically necessary

Chemotherapy:

* No prior chemotherapy for breast cancer

Endocrine therapy:

* No prior hormonal therapy for breast cancer
* No concurrent hormone replacement therapy
* No concurrent selective estrogen-receptor modulators (e.g., raloxifene for the treatment or prevention of osteoporosis)
* No concurrent oral contraceptives (i.e., birth control pills)
* No other concurrent aromatase inhibitors

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for breast cancer

Surgery:

* See Disease Characteristics
* No more than 12 weeks since prior total or partial mastectomy (including re-excision of margins)

Other:

* At least 30 days since prior investigational drugs
* No other concurrent investigational drugs
* Concurrent bisphosphonates for the treatment or prevention of osteoporosis allowed

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2104 (Actual)
Dates: Start 2000-12-04 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2014-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Levine, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Edith A. Perez, MD, Study Chair — Mayo Clinic; Kathy S. Albain, MD, Study Chair — Loyola University; Margot Burnell, Study Chair — Atlantic Health Sciences Corporation, Saint John NB; Hope Rugo, Study Chair — Cancer and Leukemia Group B
Locations (78):
- United States (44):
  - Sparks-Arkansas Oklahoma Cancer Treatment Centre, Fort Smith, Arkansas
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Scripps Cancer Center, La Jolla, California
  - University of Colorado Cancer Centre, Aurora, Colorado
  - Greenwich Hospital - Bendheim Cancer Center, Greenwich, Connecticut
  - Sibley Memorial Hospital, Oncology Research, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Centre at Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Therapy Associates, Inc., Hematology/Oncology, Evansville, Indiana
  - Lexington Oncology Assts./Central Baptist Hospital, Lexington, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - CHRISTUS Schumpert Medical Center - Hem/Onc Clinic, Shreveport, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Maine General Medical Center, Waterville, Maine
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - Associates in Oncology/Hematology, Rockville, Maryland
  - Saint Joseph Medical Center, Cancer Care Program, Towson, Maryland
  - Baystate Regional Cancer Program, Springfield, Massachusetts
  - St. Luke's Cancer Care Centre, Duluth, Minnesota
  - University of Minnesota Cancer Centre, Minneapolis, Minnesota
  - Columbia-Capitol Comprehensive Care Clinics, Jefferson City, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Creighton University Cancer Centre, Omaha, Nebraska
  - Advanced Oncology Associates, Armonk, New York
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - Winthrop University Hospital Onc/Hem, Mineola, New York
  - Hematology Oncol. Associates Rockland, Nyack, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - ECU School of Medicine, Leo Jenkins Cancer Center, Greenville, North Carolina
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - Pottstown Memorial Regional Cancer Centre, Pottstown, Pennsylvania
  - Santee Hematology Oncology, Sumter, South Carolina
  - University Oncology and Hematology Associates, Chattanooga, Tennessee
  - Lone Star Oncology Consultants, PA, Austin, Texas
  - Center for Oncology Research and Treatment, Dallas, Texas
  - Northern Utah Associates, Ogden, Utah
  - Arlington-Fairfax Hematology Oncology P.C., Arlington, Virginia
- Canada (34):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - The Royal Victoria Hospital, Barrie, Ontario
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - West Toronto, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Hotel Dieu du Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burnell MJ, O'Connor EM, Chapman JW, et al.: Triple-negative receptor status and prognosis in the NCIC CTG MA.21 adjuvant breast cancer trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-550, 2008.
- [Result] Burnell MJ, Levine MN, Chapman JA, et al.: A phase III adjuvant trial of sequenced EC + filgrastim + epoetin-alpha followed by paclitaxel compared to sequenced AC followed by paclitaxel compared to CEF in women with node-positive or high-risk node-negative breast cancer (NCIC CTG MA.21). [Abstract] J Clin Oncol 25 (Suppl 18): A-550, 2007.
- [Result] Burnell M, Levine M, Chapman JA, et al.: A randomized trial of CEF versus dose dense EC followed by paclitaxel versus AC followed by paclitaxel in women with node positive or high risk node negative breast cancer, NCIC CTG MA.21: results of an interim analysis. [Abstract] 29th Annual San Antonio Breast Cancer Symposium, December 14-17, 2006, San Antonio, Texas. A-53, 2006.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: CEF | Arm 2: EC/T | Arm 3: AC/T
Started | 701 | 701 | 702
Completed (Only 2043 patients reported toxicity data.) | 680 | 688 | 675
Not Completed | 21 | 13 | 27

BASELINE CHARACTERISTICS:
Population: Intent to treatment population is used.
  One patients from arm 1 has missing baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: CEF | Arm 2: EC/T | Arm 3: AC/T | Total
Number analyzed (Participants) | 700 | 701 | 702 | 2103
Age, Continuous [Median (Full Range); unit: years] | 48.1 [23.4 to 63.8] | 47.6 [22.7 to 61.0] | 47.6 [23.5 to 61.0] | 47.7 [22.7 to 63.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 700 | 701 | 702 | 2103
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 6 | 3 | 20
  Asian | 13 | 30 | 31 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 26 | 33 | 39 | 98
  White | 633 | 624 | 609 | 1866
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 6 | 20 | 43
Performance status [Count of Participants; unit: Participants] — Performance Status:
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    0 | 588 | 588 | 590 | 1766
    1 | 109 | 113 | 109 | 331
    2 | 3 | 0 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: Disease free survival was defined as the time from randomization to the time of recurrence of the primary disease. Local or nodal recurrence and metastatic disease were considered a recurrence of the primary tumour. Patients who had contralateral breast cancer or a second primary malignancy, or died from some cause other than disease were censored as relapse-free at the time of death. Patients who had not relapsed were censored at longest follow-up or at non-breast cancer death. As required, adjudication was used to assess reports of recurrence.
Time Frame: 13 years
Population: Intent to treat population was used for this analysis,.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: CEF | Arm 2: EC/T | Arm 3: AC/T
Number analyzed (Participants) | 701 | 701 | 702
Participants
  Disease Recurrence | 141 | 135 | 191
  No recurrence | 560 | 566 | 511
Statistical Analysis 1: Comparison: Arm 1: CEF vs Arm 2: EC/T vs Arm 3: AC/T; Test type: Superiority; p = 0.0007, Log Rank

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the time of death from any cause, with censoring at longest follow-up.
Time Frame: 13 years
Population: Intention to treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: CEF | Arm 2: EC/T | Arm 3: AC/T
Number analyzed (Participants) | 701 | 701 | 702
Participants
  Death | 123 | 107 | 146
  Alive | 578 | 594 | 556
Statistical Analysis 1: Comparison: Arm 1: CEF vs Arm 2: EC/T vs Arm 3: AC/T; Test type: Superiority; p = 0.084, Log Rank

ADVERSE EVENTS:
Time Frame: 13 years
Description: Serious and Other Adverse Events were assessed in participants who received protocol treatment. All-cause mortality was collected for all enrolled participants based on intention to treat population.
Arm/Group | Arm 1: CEF | Arm 2: EC/T | Arm 3: AC/T
All-Cause Mortality (participants affected / at risk) | 123/701 | 107/701 | 146/702
Serious Adverse Events (participants affected / at risk) | 83/680 | 86/688 | 23/675
Other Adverse Events (participants affected / at risk) | 680/680 | 688/688 | 673/675
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: CEF (N=680) | Arm 2: EC/T (N=688) | Arm 3: AC/T (N=675)
Hemoglobin (Blood and lymphatic system disorders) | 11 | 15 | 0
Transfusion: Platelets (Blood and lymphatic system disorders) | 0 | 1 | 0
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 49 | 41 | 8
Edema (Cardiac disorders) | 1 | 0 | 0
Ischemia/infarction (Cardiac disorders) | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Double vision (Eye disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 2 | 0
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 3
Proctitis (Gastrointestinal disorders) | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 12 | 12 | 1
Vomiting (Gastrointestinal disorders) | 3 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Fatigue (General disorders) | 5 | 7 | 1
Rigors, chills (General disorders) | 1 | 3 | 1
Chest pain (General disorders) | 2 | 1 | 0
Pain-Other (General disorders) | 2 | 2 | 0
Injection site reaction (General disorders) | 0 | 3 | 0
Allergic reaction (Immune system disorders) | 1 | 1 | 1
Other (Immune system disorders) | 1 | 0 | 0
Fever (Immune system disorders) | 4 | 8 | 2
Other (Immune system disorders) | 0 | 1 | 0
Other (Immune system disorders) | 1 | 2 | 1
Catheter-related infect (Infections and infestations) | 0 | 1 | 0
Wound-infectious (Infections and infestations) | 0 | 1 | 1
Granulocytes (Investigations) | 18 | 16 | 4
Platelets (Investigations) | 10 | 14 | 0
Leukocytes (total WBC) (Investigations) | 7 | 9 | 0
Cardiac troponin T (Investigations) | 0 | 0 | 1
Alkaline phosphatase (Investigations) | 0 | 1 | 0
SGPT (ALT) (Investigations) | 0 | 1 | 0
SGOT (AST) (Investigations) | 1 | 1 | 0
Bilirubin (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0
Mouth dryness (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 0
CNS hemorrhage/bleed (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 2 | 1
Seizure(s) (Nervous system disorders) | 1 | 0 | 0
Vertigo (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 1
Neuropathic pain (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginitis (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Hypotension (Vascular disorders) | 3 | 1 | 0
Thrombosis/embolism (Vascular disorders) | 7 | 5 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: CEF (N=680) | Arm 2: EC/T (N=688) | Arm 3: AC/T (N=675)
Lymphedema (Blood and lymphatic system disorders) | 31 | 26 | 51
Edema (Cardiac disorders) | 112 | 108 | 110
Cardiac LVF (Cardiac disorders) | 185 | 147 | 130
Palpitations (Cardiac disorders) | 29 | 45 | 36
Blurred vision (Eye disorders) | 32 | 56 | 46
Dry eye (Eye disorders) | 67 | 80 | 81
Tearing (Eye disorders) | 122 | 186 | 145
Constipation (Gastrointestinal disorders) | 415 | 442 | 395
Diarrhea (Gastrointestinal disorders) | 321 | 400 | 273
Dysphagia (Gastrointestinal disorders) | 135 | 163 | 98
Mouth dryness (Gastrointestinal disorders) | 44 | 101 | 32
Dyspepsia/heartburn (Gastrointestinal disorders) | 278 | 242 | 207
Nausea (Gastrointestinal disorders) | 583 | 636 | 601
Proctitis (Gastrointestinal disorders) | 82 | 95 | 26
Stomatitis (Gastrointestinal disorders) | 554 | 554 | 431
Vomiting (Gastrointestinal disorders) | 369 | 499 | 353
Rectal bleeding (Gastrointestinal disorders) | 27 | 45 | 11
Abdominal pain (Gastrointestinal disorders) | 78 | 93 | 97
Rectal/perirectal pain (Gastrointestinal disorders) | 25 | 35 | 11
Fatigue (General disorders) | 643 | 649 | 621
Rigors, chills (General disorders) | 56 | 67 | 42
Chest pain (General disorders) | 37 | 51 | 36
Pain-Other (General disorders) | 151 | 198 | 171
Injection site reaction (General disorders) | 130 | 162 | 70
Fever (Immune system disorders) | 106 | 170 | 79
Infection w/o neutropen (Infections and infestations) | 181 | 234 | 162
Febrile neutropenia (Infections and infestations) | 156 | 113 | 31
Wound-infectious (Infections and infestations) | 24 | 47 | 30
Weight loss (Investigations) | 17 | 68 | 7
Anorexia (Metabolism and nutrition disorders) | 323 | 431 | 296
Dehydration (Metabolism and nutrition disorders) | 38 | 56 | 25
Muscle weakness (Musculoskeletal and connective tissue disorders) | 31 | 57 | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 241 | 497 | 457
Myalgia (Musculoskeletal and connective tissue disorders) | 262 | 521 | 500
Bone pain (Musculoskeletal and connective tissue disorders) | 100 | 235 | 122
Taste disturbance (Nervous system disorders) | 205 | 269 | 202
Dizziness (Nervous system disorders) | 218 | 265 | 185
Memory loss (Nervous system disorders) | 21 | 32 | 44
Neuropathy-motor (Nervous system disorders) | 29 | 63 | 44
Neuropathy-sensory (Nervous system disorders) | 179 | 499 | 474
Headache (Nervous system disorders) | 229 | 308 | 266
Neuropathic pain (Nervous system disorders) | 20 | 50 | 44
Anxiety (Psychiatric disorders) | 117 | 151 | 156
Insomnia (Psychiatric disorders) | 181 | 218 | 199
Depression (Psychiatric disorders) | 100 | 129 | 101
Urine frequency/urgency (Renal and urinary disorders) | 32 | 39 | 27
Vaginitis (Reproductive system and breast disorders) | 49 | 56 | 38
Irregular menses (Reproductive system and breast disorders) | 290 | 352 | 269
Vaginal dryness (Reproductive system and breast disorders) | 45 | 52 | 36
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 104 | 205 | 171
Cough (Respiratory, thoracic and mediastinal disorders) | 147 | 231 | 177
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 297 | 320 | 241
Sweating (Skin and subcutaneous tissue disorders) | 49 | 66 | 64
Alopecia (Skin and subcutaneous tissue disorders) | 635 | 641 | 636
Dry skin (Skin and subcutaneous tissue disorders) | 61 | 89 | 58
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 22 | 106 | 20
Nail changes (Skin and subcutaneous tissue disorders) | 104 | 310 | 100
Pigmentation changes (Skin and subcutaneous tissue disorders) | 23 | 52 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 35 | 43
Rash/desquamation (Skin and subcutaneous tissue disorders) | 158 | 202 | 156
Other (Skin and subcutaneous tissue disorders) | 28 | 47 | 38
Phlebitis (Vascular disorders) | 22 | 42 | 11
Thrombosis/embolism (Vascular disorders) | 52 | 46 | 11
Hot flashes/ flushes (Vascular disorders) | 435 | 467 | 470
Flushing (Vascular disorders) | 8 | 45 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No